CLINICAL TRIAL: NCT05635604
Title: Molecular Stratification of Signaling Pathways Underlying Migraine Pathophysiology.
Brief Title: Migraine Induction Properties of PACAP-38 After Eptinezumab in Migraine Without Aura Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, Study investigator, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: H22038923
Record Dates: First submitted 2022-11-15; First posted 2022-12-02 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Migraine
Keywords: Headache; Vascular effect
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — eptinezumab; Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled design in migraine without aura patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eptinezumab and PACAP-38 (Active Comparator): The participants will receive an intravenous infusion of eptinezumab (300 mg) over 30 minutes followed (2 hours later) by an intravenous infusion of PACAP-38 (10 pmol/kg/min) over 20 minutes.
  Interventions: Drug: Eptinezumab; Drug: PACAP-38
- Placebo and PACAP-38 (Placebo Comparator): The participants will receive an intravenous infusion of placebo (saline) over 30 minutes followed (2 hours later) by an intravenous infusion of PACAP-38 (10 pmol/kg/min) over 20 minutes.
  Interventions: Drug: PACAP-38

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab or ALD403 is a humanized anti-calcitonin gene-related peptide IgG1 monoclonal antibody that binds to calcitonin gene-related peptide (CGRP). It selectively binds human CGRP ligand to prevent activation of the CGRP receptor and blocks its binding to the receptor for the prevention of migraine.
  Arms: Eptinezumab and PACAP-38
Drug: PACAP-38 — PACAP-38 is a naturally occurring peptide diffusely expressed throughout the body. The Danish Headache Center has used infusion of PACAP-38 for several years and the first time in 2007 where infusion of PACAP-38 triggered headaches and migraines in migraine patients.

SUMMARY:
To investigate whether administration of calcitonin gene-related peptide (CGRP) binding monoclonal antibodies eptinezumab prevents pituitary adenylate cyclase-activating polypeptide-38 (PACAP-38) induced migraine attacks in migraine without aura patients.

DETAILED DESCRIPTION:
The aim of the present study is to investigate whether

- CGRP binding monoclonal antibodies eptinezumab prevents PACAP-38 induced migraine attacks in migraine without aura patients.

Clinical and basic research have established calcitonin gene-related peptide (CGRP) as central molecule in migraine pathophysiology, yet existing CGRP antagonizing therapies such as the CGRP and CGRP receptor binding monoclonal antibodies are only effective in 50-60% of migraine patients. PACAP-38 and CGRP colocalize in the trigeminovascular system, and both activate adenylate cyclase upon receptor binding which causes increased formation of cyclic AMP (cAMP). It is unknown if CGRP and PACAP-38 signaling pathways differ sufficiently for PACAP-38 to be an alternative treatment target to CGRP. Whether administration of CGRP binding monoclonal antibodies eptinezumab prevents PACAP-38 induced migraine attacks in migraine without aura patients is yet to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes.
* 18-60 years.
* 50-100 kg.
* Women of childbearing potential must use adequate contraception
* History of migraine without aura for ≥ 12 months according to the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria.
* No migraine preventive treatment.

Exclusion Criteria:

* A history of serious somatic disease
* > 50 years of age at migraine onset.
* History of any other primary headaches disorder (except ≤ 5 monthly days with tension- type headache).
* Daily intake of any medication except contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
A subjective report of a migraine attack | Time of reporting migraine attack is from the baseline to 24 hours after eptinezumab/placebo administration.
  The participants report whether they feel a migraine attack (Yes or no).

SECONDARY OUTCOMES:
Headache | Time of headache measurements is from from the baseline to 24 hours eptinezumab/placebo administration.
  Headache intensity will be recorded by numerical rating scale (NRS) from 0 to 10 (0, no headache; 1, a feeling of pressure; 10, worst imaginable headache).
Changes in the superficial temporal artery (STA). | Time of headache measurements is from from the baseline to 24 hours eptinezumab/placebo administration.
  Diameter of the frontal branch of the superficial temporal artery (STA).
  Repeated measurements covering the diameter of STA before and after eptinezumab/placebo administration and PACAP-38 infusion measured by millimeters (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Danish headache center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Karagholi MA, Zhuang ZA, Beich S, Ashina H, Ashina M. PACAP38-induced migraine attacks are independent of CGRP signaling: a randomized controlled trial. J Headache Pain. 2025 Apr 14;26(1):79. doi: 10.1186/s10194-025-02022-2. PMID 40229719